CLINICAL TRIAL: NCT03960320
Title: Health Related Quality of Life of Patients With Abdominal Wall Defects
Status: Completed | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: CK-001
Record Dates: First submitted 2019-05-13; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Quality of Life; Abdominal Wall Defect; Gastroschisis; Omphalocele
Keywords: KINDL; SDQ; SF-36
MeSH Terms: conditions — Gastroschisis; Hernia, Umbilical | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire to assess the quality of life of children using KINDL, SDQ and SF-36

SUMMARY:
Examination of the health-related quality of life of patients operated on due to congenital defects of the abdominal wall after birth with the questionnaires KINDL, SDQ and SF-36.

DETAILED DESCRIPTION:
Data of all patients with a congenital abdominal wall defect (CAWD) undergoing surgical repair between 1996 and 2011 in the Department of Pediatric Surgery of the Clinic for General Surgery, Visceral, Vascular and Pediatric Surgery of the Saarland University Medical Center in Homburg were retrieved from surgical health records. Up to 2001 these records were paper based and later on electronically available (SAP enhancement package 7 for SAP ERP 6.0: 2013, Walldorf, Germany). Except epidemiological data the type of disease, data concerning birth details, pre- and postnatal course, treatment, weight and growth development have been collected electronically.

Gastroschisis or omphalocele can be simple or complex. The investigators defined complex as involvement of stenosis, atresia, ischemia, volvulus or perforation, closed or vanishing gastroschisis, and chromosomal anomalies. Giant omphalocele was considered as complex as well. The type of the primary operative procedure, primary closure of the defect or other (patch plastic etc.), was also noted. The implementation of silo technique with delayed primary closure was regarded as primary closure.

A prospective analysis was conducted by a survey with age-related questionnaires to investigate the patient´s HrQoL. The study protocol was approved by the ethical board of Aerztekammer of Saarland (Nr. 206/2013). Informed consent was given by all participating patients or their guardians.

The data collection was carried out by telephone interview, personal interview or by regular mail. The interview was always conducted by the same person, a medical student (KK). The data was collected using age related questionnaires. Together with the collection of clinical data the investigators used the validated questionnaires KINDL, SDQ and SF-36.

The KINDL questionnaire (www.KINDL.org) is a specifically developed questionnaire for children, which was developed to assess the HrQoL of life of children and adolescents. The reference values were published as part of the study "The Children and Youth Health Survey (KIGGS)" by the Robert Koch Institute, Berlin, Germany and covers the health data of 17.641 children and adolescents in Germany aged 0-17 years.

The SDQ (Strengths and Difficulties Questionnaire) is the second questionnaire that was used. The investigators used the Woerner adjustment of the SDQ as it was transferred to a German cohort.

Since there are also some adult patients in the patient collective, the investigators have also integrated the SF-36, which was developed for adolescents and adult patients.

The SF-36 is an internationally recognized and widely used questionnaire for the assessment of health-related quality of life. It records eight different dimensions (= subscales) of quality of life: physical functioning, physical role function, pain, general health perception, vitality, social functioning, emotional role function and psychological well-being. Additionally, the overall physical sum score and overall psychological sum score are listed. German reference values are available as a reference for the SF-36.

In addition, disease specific questions were asked. These included somatic and clinical data about gastrointestinal function, cosmetic aspects and scars, problems during pregnancy of the child, actual clinical health status and psycho-social development. Answers were given as precise numbers or rated according to the following LIKERT-scale with these possibilities "never-seldom-sometimes-often-always".

All data were collected and processed in an Excel spreadsheet (Microsoft® Excel®, Microsoft Corporation, Redmond, Washington, USA). The statistical analysis was carried out with SPSS (IBM® SPSS® Statistics, Version 25, International Business Machines Corporation (IBM), Armonk, New York, USA) and Excel as well.

ELIGIBILITY:
Inclusion Criteria:

* Congenital abdominal wall defect
* Surgically corrected in our department
* Survivor

Exclusion Criteria:

* Not surgically corrected in our department
* Non-Survivor

Ages: 1 Day to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with congenital abdominal wall defect, e.g. gastroschisis or omphalocele
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Differences of Kindl test results of participants with congenital wall defects compared to a norm sample of German healthy children | Day 1. For one participant all of the questionnaires were administered in one day and for that participant the study lasted one day.
  Kindl test for measuring the quality of life of participants with congenital wall defects compared to a norm sample of German healthy children
Differences of SDQ test results of participants with congenital wall defects compared to a norm sample of German healthy children | Day 1. For one participant all of the questionnaires were administered in one day and for that participant the study lasted one day.
  SDQ test for measuring the quality of life of participants with congenital wall defects compared to a norm sample of German healthy children
Differences of SF-36 results of participants with congenital wall defects compared to a norm sample of German healthy adults | Day 1. For one participant all of the questionnaires were administered in one day and for that participant the study lasted one day.
  SF-36 test for measuring the quality of life of participants with congenital wall defects compared to a norm sample of German healthy adults

CONTACTS AND LOCATIONS:
Overall Officials: Clemens-Magnus Meier, MD, Principal Investigator — Universität des Saarlandes

IPD SHARING:
Plan to Share IPD: Undecided
The publication of the data in anonymous form is planned.